CLINICAL TRIAL: NCT01167556
Title: Motivational Interviewing and Interaction Skills Training for Carers to Change Cannabis Use in Young Adults With Recent-onset Schizophrenia: Randomised Controlled Trial
Brief Title: Family Motivational Intervention in Schizophrenia
Acronym: FMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Don Linszen/ MD, PhD, AMC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Grant 100003014
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2008-02

CONDITIONS: Cannabis; Schizophrenia
Keywords: Family intervention; Recent-onset schizophrenia; Motivational Interviewing; Cannabis use
MeSH Terms: conditions — Marijuana Abuse; Schizophrenia

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Family Motivational Intervention (Experimental): An intervention provided to parents consisting of 6 sessions of training in Interactions Skills and 6 sessions training in Motivational Interviewing.
  Interventions: Behavioral: Family Motivational Intervention
- Routine care for parents (Active Comparator): Routine care for parents consisting of 2 sessions psycho-education and individual support
  Interventions: Behavioral: Family Motivational Intervention

INTERVENTIONS:
Behavioral: Family Motivational Intervention — A intervention with provided parents 6 sessions of Interaction Skills training and 6 sessions Motivational Interviewing training.

SUMMARY:
Cannabis use by people with schizophrenia is associated with family distress and poor clinical outcomes. Therefore, an Family Motivational Intervention (FMI) was developed to help parents to motivate their child with a diagnoses of recent-onset schizophrenia to reduce cannabis use.

In a single-blind randomised clinical trail with 75 patients with the diagnosis of schizophrenia, parents will be assigned to either FMI or to routine care. Assessments will be conducted at baseline and at a 10- and 22-month follow-up. The study hypothesis is that FMI will be more effective than routine care in reducing (a) cannabis use in patients and (b) distress and sense of burden in parents.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or psychotic-related disorder
* Onset of schizophrenia or related disorder within pervious the 10 years
* Cannabis use at least 2 days per week in the 3 months prior to the assessment
* Antipsychotic medication in prescribed or indicated
* At least 10 hours of contact with the parents each week in the last month

Exclusion Criteria:

-

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2006-03; Primary Completion 2010-08 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Cannabis use in patients with a diagnosis of recent-onset schizophrenia | Baseline (before the start of the intervention)
Cannabis use in patients with a diagnosis of recent-onset schizophrenia | 10-month follow-up (3 months after the intervention has ended)
Cannabis use in patients with a diagnosis of recent-onset schizophrenia | 22-month follow-up (15 months after the intervention has ended)

SECONDARY OUTCOMES:
Medication adherence in patients with a diagnosis of recent-onset schizophrenia | Baseline (before the start of the intervention)
Medication adherence in patients with a diagnosis of recent-onset schizophrenia | 10-month follow-up (3 months after the intervention has ended)
Medication adherence in patients with a diagnosis of recent-onset schizophrenia | 22-month follow-up (15 months after the intervention has ended)
Quality of life in patients with recent-onset schizophrenia | Baseline (before the start of the intervention)
Quality of life in patients with recent-onset schizophrenia | 10-month follow-up (3 months after the intervention has ended)
Quality of life in patients with recent-onset schizophrenia | 22-month follow-up (15 months after the intervention has ended)
Stress in parents due to caring for a child with recent-onset schizophrenia | Baseline (before the start of the intervention)
Stress in parents due to caring for a child with recent-onset schizophrenia | 10-month follow-up (3 months after the intervention has ended)
Stress in parents due to caring for a child with recent-onset schizophrenia | 22-month follow-up (15 months after the intervention has ended)
Expressed emotion in parents of patients with recent-onset schizophrenia | Baseline (before the start of the intervention)
Expressed emotion in parents of patients with recent-onset schizophrenia | 10-month follow-up (3 months after the intervention has ended)
Expressed emotion in parents of patients with recent-onset schizophrenia | 22-month follow-up (15 months after the intervention has ended)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Schippers, Prof. dr., Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Don Linszen, Prof.dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Lieuwe de Haan, Dr., Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Dekker N, Smeerdijk AM, Wiers RW, Duits JH, van Gelder G, Houben K, Schippers G, Linszen DH, de Haan L. Implicit and explicit affective associations towards cannabis use in patients with recent-onset schizophrenia and healthy controls. Psychol Med. 2010 Aug;40(8):1325-36. doi: 10.1017/S0033291709991814. Epub 2009 Nov 17. PMID 19917142